CLINICAL TRIAL: NCT01573091
Title: Cardiac Resynchronization Therapy Modular Registry
Acronym: CRT-MORE
Status: Completed | Type: Observational
Sponsor: Giuseppe Ricciardi (Other)
Responsible Party: Sponsor-Investigator, Giuseppe Ricciardi, Principal Investigator, University of Florence
Organization: University of Florence (Other)
Other Study IDs: 2011/0043537
Record Dates: First submitted 2012-04-02; First posted 2012-04-06 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronization therapy; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Heart failure patients: Patients with a CRT device according to current guidelines
  Interventions: Procedure: Cardiac Resynchronization Therapy

INTERVENTIONS:
Procedure: Cardiac Resynchronization Therapy — Any commercially available Cardiac Resynchronization Therapy devices with or without defibrillation backup (CRT-D/CRT-P) can be used upon discretion of the investigator according to current guidelines

SUMMARY:
The purpose of the study is to collect some parameters (clinical, electrical, radiographic, echocardiographic and ECG) able to predict response to cardiac resynchronization therapy.

DETAILED DESCRIPTION:
Heart failure is a complex clinical syndrome characterized by a high prevalence and incidence in populations at greatest risk and, therefore, with a significant social and economic impact. Randomized clinical trials, meta-analyzes, observational studies and controlled trials clearly demonstrated that the neuro-hormonal therapy is highly effective in reducing mortality, hospitalization and improving quality of life. In recent years the electrical therapy is playing an increasingly important role in the treatment of patients with chronic heart failure. Such importance is mainly due to the possibility of preventing sudden cardiac death by implanting an ICD and to correct the deleterious effects of electrical dyssynchrony and / or left ventricular mechanics by CRT. The CRT has proven an effective tool in reducing mortality, reducing symptoms and improving quality of life in patients already receiving optimal medical therapy. Despite the undoubted benefits that the electrical treatment has added to conventional medical therapy, a high percentage of patients does not benefit in terms of clinical and echocardiographic. The identification of non-responders to CRT is crucial in order not to submit the patients to an unnecessary and costly device whose electrical therapy proves to be ineffective. The reason for lack of response is still unclear but factors such as lead placement, device-settings and the degree of dyssynchrony before implant seems to be important. The purpose of the study is to collect some parameters (clinical, electrical, radiographic, echocardiographic and ECG) able to predict response to cardiac resynchronization therapy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic symptomatic HF despite stable, optimal drug therapy
* Indication for a cardiac resynchronisation device with or without defibrillator backup according to current guidelines
* Patients implanted with cardiac resynchronization device

Exclusion Criteria:

* Patients participating in other studies that clearly impact the clinical practice of the center
* Patients who are unable to provide informed consent
* Patients who can not perform follow-up in the center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for CRT device implanted according to current guidelines
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical response | 24 months
  Improvement in functional class status by at least one NYHA Class or remain in functional class II
Echocardiographic response of absolute increase of ≥5% in LVEF | 24 months
  Patients at follow-up to 6-12 months show an increase of the absolute value of the LVEF than 5%
Echocardiographic response of ≥15% reduction in LVESV | 24 months
  Patients at follow-up to 6-12 months show a systolic volume (LVESV) reduction greater than 15%

SECONDARY OUTCOMES:
LV lead/RV lead geometric distance | 12 months
  To investigate the correlation of LV lead/RV lead geometric distance (as measured by fluoroscopy) and reverse remodeling in cardiac resynchronization therapy (as measured by echocardiography as defined in primary outcome measure) at 12 months. The relation with LVESVi change between baseline and 12 months will be analyzed.
Change from baseline in R wave in 12-lead ECG at 12 months | 12 months
  To investigate the relationship between the ECG characteristics at baseline and response to cardiac resynchronization therapy (as measured by echocardiography as defined in primary outcome measure) at 12 months. The purpose of this objective is to evaluate the R wave in 12-lead ECG during BIV, RV and LV pacing and change from baseline at 12 months.
Number of ventricular arrhythmias after cardiac resynchronization therapy | 24 months
  To investigate the relationship between LV pacing and the number of ventricular tachycardia/fibrillation and/or appropriate/inappropriate shocks. The number and type of arrhythmia before and after upgrading to CRT device at 24 months will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Padeletti, MD, Study Chair — Department of Heart and Vessels, University of Florence, Florence, Italy.
Locations (12):
- Italy (12):
  - Ospedale Degli Infermi, Biella, Biella
  - San Giacomo e Cristoforo, Massa, Massa
  - Azienda Ospedaliera di Padova, Padua, Padova
  - Azienda Ospedaliera San Salvatore, Pesaro, Pesaro
  - Cardiovascular Department, Electrophysiology Unit, Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Department of Heart and Vessels, University of Florence, Florence
  - Department of Cardiology and Coronary Care Unit, Azienda Ospedaliera S. Antonio Abate, Gallarate
  - Department of Cardio, Thoracic and Vascular, Azienda Ospedaliera Carlo Poma, Mantova
  - Department of Heart, Electrophysiology, Clinica Mediterranea, Naples
  - Azienda Ospedale dei Colli - Monaldi, Napoli
  - Policlinico Federico II, Napoli
  - Department of Cardiology, Ospedale Civile "Misericordia e Dolce", Prato

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertaglia E, Reggiani A, Palmisano P, D'Onofrio A, De Simone A, Caico SI, Pecora D, Arena G, Marini M, Ricciardi G, Badolati S, Spotti A, Solimene F, Ferraro A, Migliore F, Botto GL, Malacrida M, Stabile G. The stricter criteria for Class I CRT indication suggested by the 2016 ESC Guidelines reliably exclude patients with a worse prognosis in comparison with the 2013 ESC indication criteria. Int J Cardiol. 2018 Dec 15;273:162-167. doi: 10.1016/j.ijcard.2018.09.027. Epub 2018 Sep 8. PMID 30217421
- [Derived] Stabile G, Pepi P, Palmisano P, D'Onofrio A, De Simone A, Caico SI, Pecora D, Rapacciuolo A, Arena G, Marini M, Pieragnoli P, Badolati S, Savarese G, Maglia G, Iuliano A, Botto GL, Malacrida M, Bertaglia E. Adherence to 2016 European Society of Cardiology guidelines predicts outcome in a large real-world population of heart failure patients requiring cardiac resynchronization therapy. Heart Rhythm. 2018 Nov;15(11):1675-1682. doi: 10.1016/j.hrthm.2018.04.011. Epub 2018 Apr 14. PMID 29665405
- [Derived] Stabile G, D'Onofrio A, Pepi P, De Simone A, Santamaria M, Caico SI, Rapacciuolo A, Padeletti L, Pecora D, Giovannini T, Arena G, Spotti A, Iuliano A, Bertaglia E, Malacrida M, Botto GL. Interlead anatomic and electrical distance predict outcome in CRT patients. Heart Rhythm. 2015 Nov;12(11):2221-9. doi: 10.1016/j.hrthm.2015.05.020. Epub 2015 May 19. PMID 26001509